CLINICAL TRIAL: NCT02114047
Title: Evaluation of Pulmonary Perfusion Heterogeneity in Patients With Chronic Thromboembolic Pulmonary Hypertension Using Functional PET Imaging
Brief Title: Pulmonary Perfusion Heterogeneity in Patients With CTEPH Using Functional PET Imaging
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Robert Scott Harris, M.D., Associate Physician, Massachusetts General Hospital
Other Study IDs: 2013D002300
Record Dates: First submitted 2014-04-02; First posted 2014-04-15 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study with evaluate blood flow in the lungs of patients prior to and after surgery for treatment.

DETAILED DESCRIPTION:
Specifically, we will evaluate the length-scale or size of blood flow alterations using filtering techniques with the objective of identifying the size of blood vessels that are obstructed by clot (large vessels versus small vessels).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is diagnosed with chronic thromboembolic pulmonary hypertension (WHO Group IV) and planning to undergo pulmonary thromboendarterectomy.
2. Subject is male or female aged > or =18 years of age and < or = 70 years.
3. Subject has undergone RHC within six months of entering the study.
4. The subject is capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
5. A signed and dated written informed consent is obtained from the subject.
6. Available to complete the study.
7. Able to lie flat and able to perform a 30 second breath hold.

Exclusion Criteria:

1. FEV1 and/or TLC < 70% predicted.
2. Inability to perform the study (by primary MD or investigator assessment).
3. Inability to perform the respiratory maneuvers necessary for the exam.
4. Subjects who have a past or present disease, which as judged by the Investigators may affect the outcome of this study.
5. The subject has suspected history of drugs or alcohol abuse within the six months prior to the screening visit.
6. The subject is a woman of childbearing potential who is pregnant, seeking to become pregnant, or has a positive pregnancy test.
7. Subject with clinical instability in the judgment of the investigator, with a heart rate > 120 bpm, respiratory rate > 24, SpO2 < 88%, blood pressure < 90/60 or > 140/90 or fever > 101, or subjects with hospitalization for progression of pulmonary hypertension or right heart failure in the three months prior to the study.
8. Subject with diagnosis of active tuberculosis, lung cancer, clinically overt bronchiectasis, allergic rhinitis, asthma, heart failure, ischemic heart disease, or COPD.
9. Subject that had a respiratory tract infection in the 4 weeks prior to the screening visit and throughout the duration of the study.
10. The subject has been exposed to a radiation dose over the past year that, when added to the radiation dose expected in this study, would exceed permissible yearly exposure as determined by the MGH radiation safety committee.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic thromboembolic pulmonary hypertension
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-02; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
perfusion heterogeneity | 4 months
  We will use a method to analyze the length-scale of perfusion heterogeneity before and after surgery for CTEPH. Briefly, this method consists of filtering the images with filters of different spatial size (length, mm) and measuring the coefficient of variation (CV) of perfusion in the imaged field. We then bin the CV into the following intervals: 12-36 mm, 36-60 mm, 60-84 mm, 84-108 mm and >108 mm and compare the CV in each bin among subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Harris, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Since imaging data can be identifying, researchers will need to write to the investigators and submit to IRB review if they would like to obtain raw imaging data.